CLINICAL TRIAL: NCT04072419
Title: Application of Enhanced Recovery After Surgery for Congenital Esophageal Atresia During Perioperative Period
Acronym: ERASforCEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, He Qiuming, Department of Neonatal Surgery of vice director doctor, Guangzhou Women and Children's Medical Center
Other Study IDs: GuangzhouWCMC123
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Atresia; Enhanced Recovery After Surgery
Keywords: esophageal atresia; enhanced recovery after surgery; perioperative management
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- enhanced recovery after surgery group: 1. weaning mechanical ventilation after surgery (less than 48h),
  2. no post-operative chest tube and urinary catheterization)
  3. Establishment of early feeding (D3 post-operative)
- control group: 1. the time of mechanical ventilation after surgery is more than 48 hours
  2. routine postoperative indwelling chest tube and urinary catheterization)
  3. Establishment of feeding after D3 post-operative

SUMMARY:
The purpose of this prospective cohort study is to evaluate the safety and effectiveness of enhanced recovery after surgery (ERAS) to perform routine thoracoscopic repair for elective esophageal atresia type C

DETAILED DESCRIPTION:
The concept of enhanced recovery after surgery was introduced by Kelhet et al. in the 1990s for colorectal surgery, and it referred to a group of measures performed during a patient's treatment course to improve operative outcomes, reduce complications, and speed up patient recovery. It is now widely applied in many surgical fields, such as thoracic surgery The esophageal atresia is a group of birth defects including a break in continuity of the esophagus with or without persistent communication with the trachea (tracheoesophageal fistula), and occurs in approximately 1 in 3500-4500 births. Refinements in surgical technique and perioperative care have dramatically decreased mortality rates of infants with EA/TEF, such that mortality is generally related to associated anomalies. Accordingly, the current focus in optimizing patient outcomes has shifted toward decreasing morbidity, including minimizing postoperative complications, speeding up recovery. One of the milestones in recent years is the introduction and rapid development of video-assisted thoracoscopic surgery (VATS). This surgical method has beneficial effects on patient's post-operative recovery and functional status without compromising surgical resection. A range of operations can now be safely performed via VATS.

Although the survival rate of EA is more than 90 percent, there are still many postoperative complications, including anastomotic leakage, recurrence of esophagotracheal fistula, esophageal stenosis, gastroesophageal reflux and other problems, which seriously affect the prognosis. For decades, in order to reduce the complications, post-operative muscle paralysis, mechanical ventilation and urinary catheterization were performed for at least 2 days as convention perioperative management. However, complications after general anesthesia and endotracheal intubation are not negligible, and urinary catheterization is associated with urethral trauma, discomfort, infection. The main reason for placement of chest tube is for post-operative monitoring. However, a chest drain is a recognized cause of post-operative pain and can affect patient's post-operative morbility as well as effective chest physiotherapy.

The current project aims to explored the possibility of ERAS approach (i.e. weaning mechanical ventilation after surgery (less than 48h), no post-operative chest tube and urinary catheterization) for specific Type C EA (the distance of blind end is less than 2.5cm, weight>2.4Kg, without related malformations (heart, kidney, for example), and without structural heart disease (excluding patent ductus arteriosus, patent foramen ovale, or atrial septal defect)).

ELIGIBILITY:
Inclusion Criteria:

1. congenital esophageal atresia with type C
2. the distance of blind end is less than 2.5cm
3. weight>2.4Kg
4. without related malformations (heart, kidney),
5. without structural heart disease (excluding patent ductus arteriosus, patent foramen ovale, or atrial septal defect)

Exclusion Criteria:

1. Type A/B/D/E esophageal atresia
2. the distance of blind end is more than 2.5cm
3. weight is less than 2.4Kg
4. with Inherited chromosomal related diseases
5. with congenital heart disease (excluding patent ductus arteriosus, patent foramen ovale, or atrial septal defect)
6. preoperative severe pneumonia need mechanical ventilation

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes congenital esophageal atresia with type C present to Guangzhou Women and Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-operative anastomotic leak | one month after surgery
  Comparison of the morbidity of anastomotic leak between ERAS group and control group, including major and minor leaks
Number of participants with post-operative recurrent fistula | two years after surgery
  Comparison of the morbidity of recurrent fistula between ERAS group and control group
Number of participants with post-operative anastomotic strictures | two years after surgery
  Comparison of the morbidity of anastomotic strictures between ERAS group and control. Anastomotic strictures defined as there are symptoms which require intervention.
Total number of participants with post-operative complications | two years after surgery
  Vocal cord dysfunction, Surgical site infection, Chylothorax, Gastroesophageal reflux, pleural effusion and other complications

SECONDARY OUTCOMES:
length of stay | up to 24 weeks
  length of hospital stay
Length of nutritional support in hospital | up to 24 weeks
  Length of nutritional support in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's Medical Cente, Guangzhou, China